CLINICAL TRIAL: NCT03777319
Title: A Randomized Open Label Trial of Spironolactone Versus Prednisolone in Corticosteroid-naïve Boys With DMD
Brief Title: Spironolactone Versus Prednisolone in DMD
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Inability to recruit participants.
Sponsor: Kevin Flanigan (Other)
Collaborators: Muscular Dystrophy Association (Other)
Responsible Party: Sponsor-Investigator, Kevin Flanigan, Professor of Neurology, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB17-00240
Record Dates: First submitted 2018-12-10; First posted 2018-12-17 (Actual); Results first posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Muscular Dystrophy, Duchenne
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Spironolactone; Prednisolone

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to either to the spironolactone treatment group or to the standard clinical dose of corticosteroids.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Spironolactone (Experimental): An anticipated twelve subjects will be prescribed a standard clinical dose of spironolactone of 1 mg/kg/day. The spironolactone will be provided as suspension.
  Interventions: Drug: Spironolactone
- Prednisolone (Active Comparator): An anticipated twelve subjects will be prescribed a standard clinical dose of prednisolone of 0.75 mg/kg/day or weekend dosing per sites standard of care. The prednisolone will be provided will be provided as suspension.
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Spironolactone — Spironolactone will be prescribed for 6 months, after which the family and primary care physician will determine to either remain on spironolactone or transfer to prednisolone.
  Arms: Spironolactone
Drug: Prednisolone — Prednisolone will be prescribed for 6 months as the clinical standard of care.
  Arms: Prednisolone

SUMMARY:
This is a randomized, open-label, pilot clinical trial of spironolactone suspension versus oral prednisolone for use in Duchenne muscular dystrophy. The goals are to determine the safety of 6 months of treatment with spironolactone treatment int he steroid-naive DMD population as well as to determine if either spironolactone or a standard clinical dose of corticosteroids results in equivalent improvement in time to complete the 100 meter timed test (100M).

DETAILED DESCRIPTION:
Until recently, the only treatment shown to improve strength and preserve ambulation in DMD patients was the use of glucocorticoids, which are accompanied by significant side effects including obesity, cushingoid features, osteoporosis, and behavioral disturbances. Spironolactone is an aldosterone antagonist primarily used as a potassium sparing diuretic that is widely used in the pediatric population, with limited side-effects including gynecomastia and hyperkalemia. Recent studies by Dr. Rafael-Fortney have evaluated the effect of spironolactone treatment in several different mouse models of DMD. Her results show that treatment of these mice demonstrates increased muscle membrane stabilization while reducing the negative side-effects typically associated with standard of care glucocorticoids. This pilot study is designed to determine whether this commonly used medication, spironolactone, may have similar beneficial effects with a lower side effect profile and be applicable to a wider population of DMD patients.

The hypothesis for this controlled pilot trial is that spironolactone and prednisolone are of equal efficacy in improving skeletal muscle function over a 6-month period, and that spironolactone will be well tolerated in this patient population.

One outcome is that both drugs demonstrate equal efficacy in motor function. This would then serve as pilot data for a longer term study.

ELIGIBILITY:
Inclusion Criteria:

* Duchenne muscular dystrophy (DMD) patients ≥4 to ≤7 years of age
* Clinical features of DMD that include proximal predominant weakness and/or gait disturbance
* Presence of a truncating mutation of the DMD gene in the patient or an affected male relative OR a muscle biopsy that demonstrates <5% dystrophin in the patient or an affected male relative
* Normal left ventricular ejection fraction by screening echocardiogram
* Ability to cooperate for testing
* No prior treatment with glucocorticoids or vamorolone
* No concomitant experimental therapies

Exclusion Criteria:

* Subject amenable to or currently being treated with eteplirsen, casimersen, or viltolarsen
* Hyperkalemia at screening
* History of or ongoing renal failure (elevated creatinine, oliguria, anuria)
* Hypersensitivity to spironolactone (rash, respiratory distress, arrhythmia, numbness or tingling of extremities)
* Current treatment with an ACEi
* Severe peptic ulcer disease or recent gastrointestinal perforations

Ages: 4 Years to 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Flanigan, MD, Principal Investigator — Nationwide Children's Hospital; Megan Waldrop, MD, Principal Investigator — Nationwide Children's Hospital
Locations (4):
- United States (4):
  - University of Iowa, Iowa City, Iowa
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Background] Manzur AY, Kuntzer T, Pike M, Swan A. Glucocorticoid corticosteroids for Duchenne muscular dystrophy. Cochrane Database Syst Rev. 2008 Jan 23;(1):CD003725. doi: 10.1002/14651858.CD003725.pub3. PMID 18254031
- [Background] Buck ML. Clinical experience with spironolactone in pediatrics. Ann Pharmacother. 2005 May;39(5):823-8. doi: 10.1345/aph.1E618. Epub 2005 Apr 5. PMID 15811903
- [Background] Rafael-Fortney JA, Chimanji NS, Schill KE, Martin CD, Murray JD, Ganguly R, Stangland JE, Tran T, Xu Y, Canan BD, Mays TA, Delfin DA, Janssen PM, Raman SV. Early treatment with lisinopril and spironolactone preserves cardiac and skeletal muscle in Duchenne muscular dystrophy mice. Circulation. 2011 Aug 2;124(5):582-8. doi: 10.1161/CIRCULATIONAHA.111.031716. Epub 2011 Jul 18. PMID 21768542
- [Background] Janssen PM, Murray JD, Schill KE, Rastogi N, Schultz EJ, Tran T, Raman SV, Rafael-Fortney JA. Prednisolone attenuates improvement of cardiac and skeletal contractile function and histopathology by lisinopril and spironolactone in the mdx mouse model of Duchenne muscular dystrophy. PLoS One. 2014 Feb 13;9(2):e88360. doi: 10.1371/journal.pone.0088360. eCollection 2014. PMID 24551095
- [Background] Lowe J, Floyd KT, Rastogi N, Schultz EJ, Chadwick JA, Swager SA, Zins JG, Kadakia FK, Smart S, Gomez-Sanchez EP, Gomez-Sanchez CE, Raman SV, Janssen PM, Rafael-Fortney JA. Similar efficacy from specific and non-specific mineralocorticoid receptor antagonist treatment of muscular dystrophy mice. J Neuromuscul Dis. 2016;3(3):395-404. doi: 10.3233/JND-160173. PMID 27822449
- [Background] Chadwick JA, Hauck JS, Lowe J, Shaw JJ, Guttridge DC, Gomez-Sanchez CE, Gomez-Sanchez EP, Rafael-Fortney JA. Mineralocorticoid receptors are present in skeletal muscle and represent a potential therapeutic target. FASEB J. 2015 Nov;29(11):4544-54. doi: 10.1096/fj.15-276782. Epub 2015 Jul 15. PMID 26178166
- [Background] Chadwick JA, Swager SA, Lowe J, Welc SS, Tidball JG, Gomez-Sanchez CE, Gomez-Sanchez EP, Rafael-Fortney JA. Myeloid cells are capable of synthesizing aldosterone to exacerbate damage in muscular dystrophy. Hum Mol Genet. 2016 Dec 1;25(23):5167-5177. doi: 10.1093/hmg/ddw331. PMID 27798095
- [Background] Alfano LN, Miller NF, Berry KM, Yin H, Rolf KE, Flanigan KM, Mendell JR, Lowes LP. The 100-meter timed test: Normative data in healthy males and comparative pilot outcome data for use in Duchenne muscular dystrophy clinical trials. Neuromuscul Disord. 2017 May;27(5):452-457. doi: 10.1016/j.nmd.2017.02.007. Epub 2017 Feb 17. PMID 28279570

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Spironolactone | Prednisolone
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Spironolactone: Twelve subjects will be prescribed a standard clinical dose of spironolactone of 1 mg/kg/day. The spironolactone will be provided as suspension.
  Spironolactone: Spironolactone will be prescribed for 6 months, after which the family and primary care physician will determine to either remain on spironolactone or transfer to prednisolone.
- Prednisolone: Twelve subjects will be prescribed a standard clinical dose of prednisolone of 0.75 mg/kg/day or weekend dosing per sites standard of care. The prednisolone will be provided will be provided as suspension.
  Prednisolone: Prednisolone will be prescribed for 6 months as the clinical standard of care.
- Total: Total of all reporting groups
Arm/Group | Spironolactone | Prednisolone | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: Change in Time to Complete a 100 Meter Timed Test.
Description: The determination of whether spironolactone has similar efficacy to glucocorticoids in improving muscle strength in steroid naïve DMD patients. This will be determined by measuring the time to complete a 100 meter timed test (100M).
Time Frame: 6 months
Measure: Number; unit: sec
Arm/Group | Spironolactone | Prednisolone
Number analyzed (Participants) | 1 | 1
sec | -0.6 | -5.3

2. Primary Outcome: Safety Will be Monitored Through Regular Review of Electrolytes.
Description: Electrolytes (Sodium, Potassium, Cloride and Carbon dioxide, mmol/L) will be measured on a monthly basis following initiation of either spironolactone or prednisolone.
Time Frame: 6 months
Measure: Number; unit: mmol/L
Arm/Group | Spironolactone | Prednisolone
Number analyzed (Participants) | 1 | 1
mmol/L
  Sodium-Baseline | 142 | 140
  Sodium-Month 1 | 142 | 140
  Sodium-Month 2 | 141 | 139
  Sodium-Month 3 | 142 | 141
  Sodium-Month 4 | 139 | 139
  Sodium-Month 5 | 139 | 139
  Sodium-Month 6 | 140 | 143
  Potassium-Baseline | 4.5 | 3.8
  Potassium-Month 1 | 4.7 | 4
  Potassium-Month 2 | 4.2 | 4.5
  Potassium-Month 3 | 4.1 | 3.9
  Potassium-Month 4 | 4.5 | 4.6
  Potassium-Month 5 | 4.5 | 4.2
  Potassium-Month 6 | 4.3 | 3.9
  Chloride-Baseline | 103 | 105
  Chloride-Month 1 | 109 | 105
  Chloride-Month 2 | 107 | 104
  Chloride-Month 3 | 103 | 105
  Chloride-Month 4 | 103 | 105
  Chloride-Month 5 | 103 | 106
  Chloride-Month 6 | 101 | 105
  CO2-Baseline | 29 | 22
  CO2-Month 1 | 22 | 24
  CO2-Month 2 | 25 | 24
  CO2-Month 3 | 27 | 24
  CO2-Month 4 | 28 | 25
  CO2-Month 5 | 28 | 26
  CO2-Month 6 | 26 | 26

3. Secondary Outcome: Efficacy: Dynamometry Score
Description: Secondary outcome measures will be Dynamometry score, which is a summation of maximum voluntary isometric contraction test values for knee flexion, knee extension, elbow flexion, and elbow extension
Time Frame: 6 months
Measure: Number; unit: kg
Arm/Group | Spironolactone | Prednisolone
Number analyzed (Participants) | 1 | 1
kg
  Elbow Flexion (Right)-Baseline | 0 | 3.6
  Elbow Flexion (Left)-Baseline | 0 | 4.1
  Elbow Extension (Right)-Baseline | 0 | 5.3
  Elbow Extension (Left)-Baseline | 0 | 4.1
  Knee Flexion (Right)-Baseline | 4.1 | 3.3
  Knee Flexion (Left)-Baseline | 2.8 | 3.4
  Knee Extension (Right)-Baseline | 3.8 | 4.8
  Knee Extension (Left)-Baseline | 5.9 | 5.2
  Elbow Flexion (Right)-Month 6 | 3.1 | 2.9
  Elbow Flexion (Left)-Month 6 | 3.5 | 3.4
  Elbow Extension (Right)-Month 6 | 2.4 | 4.3
  Elbow Extension (Left)-Month 6 | 2.5 | 3.8
  Knee Flexion (Right)-Month 6 | 4.3 | 4.1
  Knee Flexion (Left)-Month 6 | 4.1 | 3.9
  Knee Extension (Right)-Month 6 | 7.2 | 6
  Knee Extension (Left)-Month 6 | 8.3 | 5.1

ADVERSE EVENTS:
Time Frame: Data was collected for each participant over a 7 month duration.
Arm/Group | Spironolactone | Prednisolone
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Spironolactone (N=1) | Prednisolone (N=1)
Viral Illness (Gastrointestinal disorders) | 1 (2) | 0 (0)
Loose Stool (Gastrointestinal disorders) | 1 (1) | 0 (0)
Muscle Cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Dental Cavity (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Full enrollment into the study was unable to be obtained.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/19/NCT03777319/Prot_SAP_000.pdf